CLINICAL TRIAL: NCT01719315
Title: Neurophysiologic Correlates of Hypersomnia: a High Density EEG Investigation
Brief Title: Neurophysiologic Correlates of Hypersomnia
Status: Completed | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Other Study IDs: 2012-0201
Record Dates: First submitted 2012-10-24; First posted 2012-11-01 (Estimated); Last update posted 2018-12-24 (Actual); Status verified 2018-12

CONDITIONS: Major Depressive Disorder; Primary Hypersomnia; Bipolar Disorder; Narcolepsy; Primary Insomnia
MeSH Terms: conditions — Depressive Disorder, Major; Idiopathic Hypersomnia; Bipolar Disorder; Narcolepsy; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (8):
- MDD with Hypersomnia: Participants with Major Depressive Disorder and co-morbid hypersomnia
  Interventions: Other: Acoustical slow wave induction
- MDD without hypersomnia: Participants with Major Depressive Disorder but without co-morbid hypersomnia
- BPAD with hypersomnia: Participants with Bipolar Affective Disorder and co-morbid hypersomnia
  Interventions: Other: Acoustical slow wave induction
- BPAD without hypersomnia: Participants with Bipolar Affective Disorder without co-morbid hypersomnia
- Primary Hypersomnia: Patients with primary hypersomnia (idiopathic hypersomnia)
  Interventions: Other: Acoustical slow wave induction
- Primary Insomnia: Patients with primary insomnia
- Narcolepsy: Subjects with narcolepsy
  Interventions: Other: Acoustical slow wave induction
- Healthy Controls: healthy participants

INTERVENTIONS:
Other: Acoustical slow wave induction — Brief tones (50 millisecond duration) at a frequency of 0.8 and 2 Hz, a rate that approximates the natural cellular oscillations of cortical neurons during sleep, will be played in blocks of 15-20 during non-rapid eye movement (NREM) sleep. Blocks of active acoustic slow wave induction will be followed by blocks of equal duration without induction, in order to make comparisons between stimulation periods (ON) and no stimulation periods (OFF). Tone intensity will be manually adjusted so as to be above an individual participant's auditory threshold during waking, but still quiet enough as not to awaken the subject from sleep. Sham slow wave induction will consist of auditory tones played prior to sleep, and during sleep of insufficient timing and intensity to alter slow wave activity.
  Groups: BPAD with hypersomnia; MDD with Hypersomnia; Narcolepsy; Primary Hypersomnia

SUMMARY:
The goal of this project is to examine the neurophysiology of hypersomnia during sleep and wakefulness, to identify biomarkers for excessive sleepiness in neuropsychiatric disorders, and pilot acoustical slow wave induction during sleep in patients with hypersomnolence, to determine if this decreases daytime sleepiness in these patients. The primary study hypotheses are that individuals with hypersomnolence will have reduced slow wave activity (SWA) during sleep and increased waking theta/alpha activity during wake in specific brain regions. A secondary hypothesis is that acoustical slow wave induction in hypersomnolent patients will increase SWA during sleep, reduce theta/alpha activity during wake, and improve subjective sleepiness.

ELIGIBILITY:
Inclusion Criteria:

* Meet Diagnostic and Statistical Manual edition IV criteria for neuropsychiatric disorders enumerated in study population description

Exclusion Criteria:

Exclusionary criteria for all subjects will include: evidence of a clinically significant sleep disorder that would cause hypersomnolence (e.g. moderate to severe obstructive sleep apnea, restless legs syndrome, shift-work sleep disorder), history of significant head trauma or loss of consciousness > 30 minutes; current smoking of more than 15 cigarettes per day; >3 caffeinated beverages per day; significant neurologic or medical illness; active drug/alcohol abuse/dependence (within 6 months of enrollment), women who are pregnant, <6 months post-partum, nursing or planning to become pregnant during the study; left-handedness (due to effects on sleep topography); and imminent risk for self-harm or suicide.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Subjects will be recruited from the greater Madison, WI area. Hypersomnolent subject groups (n=30 in each group) may include unipolar MDD with hypersomnolence, primary hypersomnia (idiopathic hypersomnia), bipolar disorder with hypersomnolence, and narcolepsy. Non-hypersomnolent comparison groups (n=30 in each group) will include: MDD without hypersomnolence, bipolar disorder without hypersomnolence, primary insomnia, and healthy controls.
Sampling Method: Non-Probability Sample
Enrollment: 76 (Actual)
Dates: Start 2012-11 (Actual); Primary Completion 2018-06 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Nocturnal Slow Wave Activity | Individual nights of sleep recorded within an average of 4 weeks of enrollment
  EEG recordings during sleep will be analyzed to assess slow wave activity in the 1-4.5Hz range.

SECONDARY OUTCOMES:
Waking theta/alpha activity | Individual days of waking EEG will be recorded within an average of 4 weeks of enrollment
  Waking EEG activity across the 1-12Hz range will be analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: David T Plante, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin-Madison, Department of Psychiatry, Madison, Wisconsin, United States